CLINICAL TRIAL: NCT03354351
Title: Mind the Heart: Best Practices for Prevention, Early Identification and Treatment of Mood and Anxiety Disorders in Men With Heart Disease
Brief Title: Comorbid Mental Disease and Heart Disease in Men
Acronym: MindTheHeart
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universite de Moncton (Other)
Collaborators: Movember Foundation (Other); New Brunswick Health Research Foundation (Other)
Responsible Party: Principal Investigator, Jalila Jbilou, Associate professor, Universite de Moncton
Other Study IDs: MindTheHeart-UMoncton-2017
Record Dates: First submitted 2017-11-16; First posted 2017-11-27 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Acute Coronary Syndrome; Depressive Disorder; Anxiety Disorders; Stress Disorders, Post-Traumatic
Keywords: Stepped-care model; Men's health; Prevention; Early treatment; Psychotherapy
MeSH Terms: conditions — Acute Coronary Syndrome; Depressive Disorder; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NB-Group: Stepped-care model comprising a hierarchy of interventions, from the least to the most intensive, matched to the cardiac man's needs. The model involves three steps: Step 1 (therapist-guided and self-guided 3-session psychoeducational program), Step 2 (Group sessions involving care partners), and Step 3 (individual or dyadic (patient and care Partner) sessions. As such, if following Step 1, the mental-health symptoms of men with HD do not sufficiently subside, as identified by the screening tests, participants will qualify for Step 2. Following Step 2, men who continue to meet criteria for a clinically significant mood, anxiety, or post-traumatic stress disorder on the screening tests (PHQ9, MRDS, DASS 21, IES-R, CIS), will be invited to receive services at Step 3.
  Interventions: Behavioral: Stepped-care model
- ON-Group: Stepped-care model where men will need to follow a sequential treatment (Step 1 (self-guided), Step 2 (Group sessions), and Step 3 (individual or couple sessions). As such, if following Step 1, the mental-health symptoms of men with HD do not sufficiently subside, as identified by the screening tests, participants will qualify for Step 2. Following Step 2, men who continue to meet criteria for a clinically significant mood, anxiety, or post-traumatic stress disorder on the screening tests (PHQ9, MRDS, DASS 21, IES-R, CIS), will be invited to receive services at Step 3.
  Interventions: Behavioral: Stepped-care model
- QC-Group: Standard Stepped-care model where men will need to follow a sequential treatment (Step 1 (self-guided), Step 2 (Group sessions), and Step 3 (individual or couple sessions). As such, if following Step 1, the mental-health symptoms of men with HD do not sufficiently subside, as identified by the screening tests, participants will qualify for Step 2. Following Step 2, men who continue to meet criteria for a clinically significant mood, anxiety, or post-traumatic stress disorder on the screening tests (PHQ9, MRDS, DASS 21, IES-R, CIS), will be invited to receive services at Step 3.
  Interventions: Behavioral: Stepped-care model

INTERVENTIONS:
Behavioral: Stepped-care model — The intervention proposed in this study is a stepped-care model (comprising 3 steps) integrating cognitive-behavioural therapy or trauma-focused therapy and emotion-focused therapy that involves matching individuals to the most appropriate level of care, based on their specific needs . When patients do not show improvement they move to higher, more intensive levels of care.
  Other Names: MindTheHeart

SUMMARY:
Mood disorders, anxiety disorders, and trauma-related stress (MD\AD\TRS) are common among men, particularly those suffering from heart disease (HD). MD\AD\TRS are significantly related to exacerbation of HD symptoms that often lead to death. Unfortunately, men are significantly less likely than women to seek and receive appropriate treatment for their mental health issues including MD\AD\TRS. Furthermore, there is little literature about the use of the stepped care model in the Canadian setting.

The overarching goal of this interventional program is therefore to prevent, early detect and treat MD\AD\TRS in men living with HD. This Participatory Action Research aims to implement a stepped-care model for MD\AD\TRS in men in New Brunswick, Ontario, and quebec. The second phase of the project proposes a quantitative study that will consist of testing the effectiveness and acceptability (by the men and the involved health professionals) of the stepped-care model. It will offer to post ACS-males a mental health related component presently not available in the typical services of the NB health system.

Data will be collected at baseline (0 month) and at four follow-up (each 3-months) sessions to manage the progress of each participant throughout their 12-month journey in the study. Typical sociodemographic data will be collected, along with a questionnaire on Masculinity Norms, Couples Satisfaction (when applicable), and four mental health assessment tools.

DETAILED DESCRIPTION:
The intervention proposed in this study is a stepped-care model comprised of three steps. The intensity of the intervention increases for participants with each of the following steps: 1) psychoeducation, 2) group therapy and 3) individual therapy. Recent evidence has shown the need for more tailored assessment and treatment methods for men suffering from depression as well as evidence showing the effectiveness of EFT (Emotionally-Focused Therapy)1. As such, the stepped-care model approach will be based on cognitive-behaviour therapy (CBT) and Emotionally-Focused Therapy (EFT). The research design is based on a quasi-experimental paradigm and a prospective observational cohort study.

Background information In 2012, the Canadian Institute for Health Information estimated that 6.8 million Canadians age 20 to 74 are affected by the following chronic conditions heart disease, high blood pressure, diabetes, asthma, and chronic obstructive pulmonary disease. Strikingly, nearly 40% more men than women are likely to be hospitalized for all types of heart disease (HD) combined2. Mental health and physical health are fundamentally linked. It is three times more likely that a person with HD will experience depression when compared to people without HD2. Research on men's mental health in the context of HD, specifically in acute coronary syndrome (ACS), reveals an important relationship between HD and mood disorders, anxiety disorders, and trauma-related stress in men (MD/AD/TRS)3. Co-existing HD and mental illness contribute to worse health status and higher health care utilization rates3. This is problematic because men underuse mental health services and health services in general4. The principal reasons evoked to explain this are the lack of "male-friendly" health services, the functional view that men have of their bodies, and their perception of healthcare services as occasional "fix-it" cures4. Thus, while men appear to be at high risk for HD and for the spectrum of MD/AD/TRS that often accompany it and slow the rehabilitation from ACS, they are unlikely to receive preventative services, to seek and to receive appropriate timely interventions for their psychological distress and mental illness. This in turn, can jeopardize men's mental health, quality of life and physical health over the long term, along with their life expectancy. Indeed, the occurrence of MD/AD/TRS has been shown to impact the prognosis of ACS patients.

In the context of this study an Acute coronary syndrome (ACS) encompasses multiple heart diseases having symptoms consistent with acute myocardial ischemia, including unstable angina and myocardial infarctions (MI) ("heart attacks") such as non-ST-segment elevation myocardial infarction (NSTEMI) and ST-segment elevation myocardial infarction (STEMI)5. On the other hand, Mood disorder or depressive disorders (MD) includes a variety of depressive conditions that mainly cause an individual to not function normally from a mental and physical standpoint. These conditions all show symptoms of sadness, emptiness and irritable mood6. Anxiety disorders (AD) consist of the anticipation of future threats, which cause an individual to be overly cautious or avoidant and result in such actions as misguided or anticipatory muscle tension in normal-considered situations6. Trauma-related stress (TRS) describes a condition where the individual's exposure to an event has caused unusual, physical or mental, stress or trauma. The aftermath of these events can vary; with some having the individual experiences anxiety and fear, but more often they will show a hedonic, dysphoric, dissociative and aggressive symptoms6.

Relevant Literature and Data The psychological effects of HD are seen at the patient level and their family (e.g. intimate partner)7-12. HD is related to decrease in sexual activity and sexual satisfaction, decrease in effective interpersonal communication, and increase in the amount and intensity of conflict in couple relationships13,14. This can be especially problematic for men, because they tend to become more intensely physiologically aroused (e.g., increase in blood pressure, cardiac reactivity, and limbic activation) for more extended periods of time during and after conflicts with their partners than do women15, which tends to lead them to shut down emotionally and to shut out their relationship partner in an attempt to re-establish psychological and physiological homeostasis16-18.Unfortunately, this type of "stonewalling"15 behaviour usually only serves to exacerbate couple conflict and leads to distressed conjugal relationships16-18. Clinically significant symptoms of depression and anxiety are known correlates of conjugal distress19-21. Furthermore, emotional isolation is also a known risk factor for the development of TRS22,23. Patients with MD/AD/TRS are at greater risk (two-fold) of major adverse cardiac events than those without24; and at risk of recurrent HD and mortality25. All of this may contribute to poorer prognosis of ACS patients with MD/AD/TRS.

Despite findings from some small-scale studies that indicate positive effects of psychotherapy and pharmacological therapy on symptoms of depression and anxiety in the context of HD26-28, the results of large controlled trials are equivocal. The Enhancing Recovery in Coronary HD Patients (ENRICHD) study investigated MD, HD, social support and CBT29-32. Their finding showed that CBT helped to reduce symptoms of depression in MI patients in short term but the benefits waned after 30 months. Similarly, the Cardiac Randomized Evaluation of Antidepressant and Psychotherapy Efficacy (CREATE) study suggested that 12 weeks of Interpersonal Therapy (IPT) did not add to the effects of clinical management on depression in cardiac patients when combined with the antidepressant citalopram33. The psychological treatments that have been used to date thus appear to be lacking for cardiac patients with depression, which emphasizes the need for the development of ones that will have the desired effects on their psychological symptoms. Aside from the handful of studies cited above, published reports of treatments/care of MD/AD/TRS in the context of HD are virtually nonexistent. Thus far, all of the research in this area has focused on generic treatments for men and women that might neglect the specific needs or tendencies of either gender in terms of mental-health treatment.

For aforementioned reasons, ensuring that men are properly informed, screened, and treated for MD/AD/TRS in the context of HD is essential. It is also imperative that the preventive approaches and the treatments they receive be tailored to their particular needs (e.g. goal-oriented focus with specific and attainable objectives)34. As previous literature pointed out, "The rationale behind the development of male sensitive approaches is that men generally have a harder time engaging in the activities germane to psychotherapy (e.g., identifying and discussing feelings, considering the intra- and interpersonal impact of one's own behaviour and that of others, showing vulnerability, asking for help) than do women, for a host of reasons related to both biology and socialization ." Men are significantly less likely than women to seek any kind of help for common mental-health problems4,36. Most of the psychological services routinely offered tend to focus predominantly on symptom-management, with little attention to the interpersonal connections that attenuate the loneliness and isolation that contribute to MD/AD/TRS. A notable exception to this is IPT mentioned earlier. Furthermore, to the investigators knowledge, IPT has not been applied to cardiac patients with MD/AD/TRS, and it appears to be less effective for patients with little or no social support or with dysfunctional conjugal relationships26. Recognition of the importance of interpersonal relationships for mental health has led a handful of clinical researchers to integrate relational components into their treatments for depression, anxiety, and comorbid HD and to test their efficacy26,33,37,38. However, there has not yet been, to the investigators knowledge, any systematic attempt to tailor and apply relationship-focused treatments to the needs of men suffering from MD/AD/TRS as they recover from HD. These include a focus on the intra- and interpersonal skills known to coincide with psychological health (e.g., awareness and integration of primary affect into daily interactions in order to meet socio-affective needs, realistic thinking, engagement in rewarding behaviours) and presentation of these skills in ways that will resonate with male patients (e.g., task-focused approach, appropriate rationale).

Stepped-care models have been applied elsewhere for MD/AD/TRS treatment with general success and acceptability. Studies have shown that the stepped-care implementation was received positively in primary care settings39. It was also shown to be effective in reducing symptoms and improving functioning among TRS patients40. According to the literature, the stepped care model has also been used with cardiac patients and was acceptable, effective and accessible41.

Clinical relevance of the project Currently, in the province of New Brunswick, there a few services offered or follow-ups available for ACS patients in relation to their mental health. Some cardiac rehabilitation centers in the province offer access to psychological services to ACS patients, but these are very limited compared to more intensive services such as stepped-care models. These services include access to information on depression and a more thorough Cardiac Wellness Program with access to a psychologist for patients who wish to pursue their rehabilitation42. In the past few decades, implementation of stepped-care models for the treatment of mood disorders have been seen globally43,44 and their adaptation deemed as cost-effective45-47.

The MD/AD/TRS stepped-care intervention proposed in this study will contribute to adopt men-sensitive interventions and preventive approaches (information/education and early detection) and to emphasize the link between HD and men's relationships and interpersonal support by means of including identified significant people in their lives for their treatment. Modifications to the stepped-care model will be integrated based on findings from the qualitative study in phase 1 of the project which encompassed focus groups with men and interviews with health professionals. Some of these modifications include utilizing language that is men sensitive, giving a choice to men as to whether they would like to include their partners in therapy and providing training for therapists on the stepped care model.

Objectives of the Phase 2 of the study Primary Objectives The primary objectives of this observational study is to assess the feasibility, acceptability and efficacy of the stepped-care model and thus to identify predictors of utilization, compliance and clinical trajectory of men following an ACS, experiencing or not a common mental illness (MD/AD/TRS).

Secondary Objectives

In addition, the study secondary objectives are:

* Improve the utilization of cardiac rehabilitation programs among men post-ACS.
* Assess changes of men perceptions towards masculinity and their relationship to their partners.
* Develop recommendations to support implementation and scaling-up the intervention in the province.

ELIGIBILITY:
Inclusion Criteria:

* New Brunswick, Ontario and Quebec sites:

  1. men with a diagnosis of ACS (Acute cardiac syndrome) : myocardial infarction such as ST-segment elevation myocardial infarction (STEMI), non-ST-segment elevation myocardial infarction (NSTEMI), or unstable angina, or angioplasty with or without a stent or coronary bypass in the last 3 months.
  2. able to speak or write in English or French
  3. with an identified treating health professional (cardiologist, family doctor or nurse practitioner).
  4. able to attend 8 weekly sessions if qualifies for step 2;
  5. available for at least one year of follow-up.
* New-Brunswick site only:

  1. Surgery patients (surgery in the last three months) will also be included (CABG, Percutaneous valve, Valve, Valve/Graft, Cardioverter (pacemaker), …)
  2. Congestive heart failure : patients with NYHA Class III or NYHA Class IV.

Exclusion Criteria:

* Abuse of any substance in the past 12 months such as alcohol, cannabis, drugs as screened by the Simple Screening Instrument for Substance Abuse;
* Self-reported personal history of psychotic disorders or bipolar disorders (i.e. schizophrenia, paranoia, personality disorders
* Recently (3 months or less) started on psychotherapy or pharmacological treatment of MD/AD/TRS.

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male inpatients of cardiology departments, clients of cardiac rehabilitation programs and patients refered by their cardiologist or family doctor.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline PHQ9 at 12 months | Baseline, 3 months, 6 months, 9 months and 12 months
  Questionnaire for Depression Scoring: Minimal depression (0-4); Mild depression (5-9); Moderate depression (10-14); Moderately severe depression (15-19); Severe depression (20-27)
Change from Baseline DASS-21 at 12 months | Baseline, 3 months, 6 months, 9 months and 12 months
  set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic nonspecific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.
Change from Baseline IES-R at 12 months | Baseline, 3 months, 6 months, 9 months and 12 months
  The IES-R is a 22-item self-report measure that assesses subjective distress caused by traumatic events.Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88) and subscale scores can also be calculated for the Intrusion, Avoidance, and Hyperarousal subscales.

SECONDARY OUTCOMES:
Change from Baseline CSI-32 at 12 months | Baseline, 3 months, 6 months, 9 months and 12 months
  A 32-item scale designed to measure one's satisfaction in a relationship. The scale has a variety of items with different response scales and formats. The authors have also specified that the scale safely be shrunk to either a 16-item format or even a 4-item format depending on a researcher's needs.
Change from Baseline CMNI-22 at 12 months | Baseline, 3 months, 6 months, 9 months and 12 months
  Conformity to Masculine Norms Inventory-Abbreviated version. Self-descriptive statements that measure individual behaviors, attitudes, and conformity to an assortment of dominant masculine norms in the United States.

OTHER OUTCOMES:
Change from Baseline GAD-7 at 12 months | Baseline, 3 months, 6 months, 9 months and 12 months
  The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
Change from Baseline MDRS-22 at 12 months | Baseline, 3 months, 6 months, 9 months and 12 months
  Male Depression Risk Scale (MDRS-22) is a 22-item measure that employs a 7-point rating scale (0 = not at all, 7 = almost always).

CONTACTS AND LOCATIONS:
Overall Officials: Jalila Jbilou, MD, PhD, Principal Investigator — Universite de Moncton

IPD SHARING:
Plan to Share IPD: No